CLINICAL TRIAL: NCT05145829
Title: Exploring an Alternative Pre-operative Sentinel Lymph Node Mapping Method Using a Magnetic Tracer and MRI for Melanoma Patients
Brief Title: Exploring an Alternative Pre-operative SLN Mapping Method Using a Magnetic Tracer and MRI for Melanoma Patients
Acronym: SCARLETT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, James van Bastelaar, Head of department of Surgery (MD, PhD), Zuyderland Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METCZ20210156
Record Dates: First submitted 2021-11-03; First posted 2021-12-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
Keywords: Magnetic tracer; Sentinel lymph node; Melanoma; MRI
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melanoma patients (Experimental): All patients will undergo lymphatic mapping with SPIO, 99mTc and PB.
  Interventions: Diagnostic Test: Diagnostic Test: Sentinel node mapping using MRI

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Sentinel node mapping using MRI — Sentinel lymph node mapping in melanoma patients using a magnetic tracer and MRI

SUMMARY:
Sentinel lymph node biopsy (SLNB) is crucial in the management of malignant melanoma treatment and is currently performed by pre-operatively inject a colloid nanomaterial labeled with Technetium (99mTc) as radioactive tracer. Intra-operatively, Patent Blue (PB) will be injected to improve the visualization of the lymphatic tract. However, current pre-operative SLN mapping technique is associated with disadvantages as radiation exposure for both patients and health care staff and logistic challenges, because of time constraints due to short half-live time of 99mTc.

Superparamagnetic iron oxide (SPIO) is a non-radioactive technique using a magnetic tracer (Magtrace® (Endomagnetics Ltd.)) to identify SLNs. Several studies showed that SPIO is non-inferior to dual tracing with 99mTc and PB in breast cancer patients. SPIO is expected to be non-inferior to dual tracing with 99mTc and PB in melanoma patients. However, further research is needed to demonstrate the use of SPIO in pre-operative MRI scanning.

The primary objective of this study is to evaluate the feasibility and diagnostic accuracy of pre-operative MRI scanning using SPIO compared to lymphoscintigraphy (LS) and single-photon emission computed tomography/computed tomography (SPECT/CT) using 99mTc for identifying SLN status in melanoma patients.

DETAILED DESCRIPTION:
Rationale: Sentinel lymph node biopsy (SLNB) is crucial in the management of malignant melanoma treatment and is currently performed by pre-operatively inject a colloid nanomaterial labeled with Technetium (99mTc) as radioactive tracer. Intra-operatively, Patent Blue (PB) will be injected to improve the visualization of the lymphatic tract. However, current pre-operative SLN mapping technique is associated with disadvantages as radiation exposure for both patients and health care staff and logistic challenges, because of time constraints due to short half-live time of 99mTc.

Superparamagnetic iron oxide (SPIO) is a non-radioactive technique using a magnetic tracer (Magtrace® (Endomagnetics Ltd.)) to identify SLNs. Several studies showed that SPIO is non-inferior to dual tracing with 99mTc and PB in breast cancer patients. SPIO is expected to be non-inferior to dual tracing with 99mTc and PB in melanoma patients. However, further research is needed to demonstrate the use of SPIO in pre-operative MRI scanning.

Objective: The primary objective of this study is to evaluate the feasibility and diagnostic accuracy of pre-operative MRI scanning using SPIO compared to lymphoscintigraphy (LS) and single-photon emission computed tomography/computed tomography (SPECT/CT) using 99mTc for identifying SLN status in melanoma patients. A secondary objective is to assess the feasibility and diagnostic accuracy of SPIO/magnetometer (Sentimag®, Endomagnetics Ltd.) in comparison with dual trace gold standard (99mTc and PB) in SLN procedures in melanoma patients.

Study design: A prospective single-arm feasibility study will be performed at the department of Surgical oncology at Zuyderland Medical Center Sittard, the Netherlands.

Study population: Adult patients (≥18 years) with primary melanoma stage I-II and an indication for wide local excision (1 cm) and SLN procedure will be included in the study.

Intervention (if applicable): All patients will undergo lymphatic mapping with a SPIO tracer (Magtrace®), 99mTc and PB.

Main study parameters/endpoints: The concordance in SLN detection rate (sensitivity and specificity) of SPIO/MRI and LS and SPECT/CT using 99mTc.

The concordance in SLN detection rate (sensitivity and specificity) of SPIO/magnetometer and the gold standard dual trace technique using 99mTc/Gamma probe and PB. Additionally, the number of post-injection (skin) reactions, complication and adverse events will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age at the time of consent;
* Histological confirmed melanoma (patient must have primary cutaneous melanoma with Breslow thickness ≥ 0.8-2.0mm with or without ulceration or <0.8mm with ulceration (pT1b - pT2b, AJCC 8th edition));
* Indication for wide local excision (margin 1 cm) and SLN procedure;
* Patients should be willing and able to provide informed consent.

Exclusion Criteria:

* Intolerance/hypersensitivity to 99mTc-nanocolloid, PB, iron or dextran compounds;
* Iron overload disease;
* Pregnant or breast-feeding women;
* Previous surrounded lymph node surgery;
* Patients with head and neck melanomas;
* Standard MRI exclusion criteria;
* Implantable (electrical) devices (e.g. pacemaker, cochlear implants, neurostimulator);
* Any other metal implants;
* Claustrophobia;
* MR-incompatible prosthetic heart valves;
* Patients who are unable or refuse to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of SPIO/MRI and LS+SPECT/CT and 99mTc to identify SLN | Before surgery (MRI scanning and scintigraphy)
  The diagnostic accuracy of SPIO/MRI and LS+SPECT/CT and 99mTc to identify SLN will be expressed as sensitivity and specificity, and positive and negative predictive values, including their 95% exact binomial confidence intervals. MRI image analyses will be performed by two independent professionals.

SECONDARY OUTCOMES:
The diagnostic accuracy of SPIO/magnetometer and PB, 99mTc and Gamma probe | During SLNB (surgery)
  The diagnostic accuracy of SPIO/magnetometer and PB, 99mTc and Gamma probe will be expressed as sensitivity and specificity, and positive and negative predictive values, including their 95% exact binomial confidence intervals .
Comparison between 99mTc injection + LS + SPECT/CT time vs SPIO injection + MRI | During SLNB (surgery)
  Time/duration of 99mTc injection + LS + SPECT/CT and time/duration of SPIO injection + MRI will be compared
Number of post-injection (skin) reactions, complication and adverse events | At 10-14 days and at 3 months after the procedure
  Descriptive only

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No